CLINICAL TRIAL: NCT05992818
Title: Comparison of DRS-R-98 (The Delirium Rating Scale--Revised-98) and 3D-CAM (3-minute Diagnostic Assessment for CAM-Confusion Assessment Method-defined Delirium) in the Assessment of Postoperative Delirium in Elderly Patients
Brief Title: Comparison of DRS-R-98 and 3D-CAM in the Assessment of Postoperative Delirium in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ozlem Turhan, Principal Investigator, Istanbul University
Other Study IDs: 2022/2132
Record Dates: First submitted 2023-08-05; First posted 2023-08-15 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Delirium
Keywords: Elderly patients; DRS-R-98(The Delirium Rating Scale--Revised-98); 3D-CAM; delirium
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: comparing DRS-R-98 (The Delirium Rating Scale--Revised-98) and 3D-CAM (3-minute diagnostic assessment for CAM-Confusion Assessment Method-defined delirium) tests to assess postoperative delirium — determine the test that is more effective and practical in the assessment of POD

SUMMARY:
Postoperative delirium (POD) is a transient and usually fully reversible altered state of consciousness that develops acutely or subacutely after surgery, characterized by widespread, daily fluctuations in brain metabolism and function. It can be seen as hyperactive (mania), hypoactive (depressive) and mixed type. It has been shown to be associated with increased morbidity, mortality, health expenditures and prolonged hospitalization in the postoperative period. In studies, the frequency of POD was found to be 17-51% in orthopedic surgery, 11-46% in cardiac surgery and 13-50% in non-cardiac surgery. There are many studies in the literature on advanced age, comorbidities (e. g; diabetes mellitus, stroke, coronary artery disease, arrhythmias), dementia, use of glasses-hearing aids, medications (anticholinergic, opioid, benzodiazepine etc. ), duration of anesthesia, type of surgery, electrolyte disturbances, perioperative bleeding, hypotension, pain and intensive care unite stay as risk factors associated with delirium. This condition, which has a multifactorial etiology, is often unrecognized, unpreventable, untreatable and leads to increased morbidity and mortality. Therefore, it is important to recognize delirium that develops in the postoperative period and to perform the necessary interventions.

There are many tests used in the diagnosis of POD. Delirium tests; it evaluates the patient under many sub-headings such as orientation, memory, attention, visual and spatial ability.

The gold standard method is DSM-V (North American Diagnostic and Statistical Manual-V of Mental Disorders-V) to assess delirium status. There are also some other tests like DRS-R-98 (The Delirium Rating Scale--Revised-98) and 3D-CAM (3-minute diagnostic assessment for CAM-Confusion Assessment Method-defined delirium). In addition to patient assessment, these tests are useful for the clinician in the diagnosis of delirium.

The aim of the study is to compare the DRS-R-98 and 3D-CAM tests used in the assessment of POD, and to evaluate their feasibility and the power detecting delirium.

DETAILED DESCRIPTION:
Postoperative delirium (POD) is a transient and usually fully reversible altered state of consciousness that develops acutely or subacutely after surgery, characterized by widespread, daily fluctuations in brain metabolism and function. It can be seen as hyperactive (mania), hypoactive (depressive) and mixed type. It has been shown to be associated with increased morbidity, mortality, health expenditures and prolonged hospitalization in the postoperative period. In studies, the frequency of POD was found to be 17-51% in orthopedic surgery, 11-46% in cardiac surgery and 13-50% in non-cardiac surgery. There are many studies in the literature on advanced age, comorbidities (e. g; diabetes mellitus, stroke, coronary artery disease, arrhythmias), dementia, use of glasses-hearing aids, medications (anticholinergic, opioid, benzodiazepine etc. ), duration of anesthesia, type of surgery, electrolyte disturbances, perioperative bleeding, hypotension, pain and intensive care unite stay as risk factors associated with delirium. This condition, which has a multifactorial etiology, is often unrecognized, unpreventable, untreatable and leads to increased morbidity and mortality. Therefore, it is important to recognize delirium that develops in the postoperative period and to perform the necessary interventions.

There are many tests used in the diagnosis of POD. Delirium tests; it evaluates the patient under many sub-headings such as orientation, memory, attention, visual and spatial ability. The gold standard method is DSM-V (North American Diagnostic and Statistical Manual-V of Mental Disorders-V) to assess delirium status. There are also some other tests like DRS-R-98 (The Delirium Rating Scale--Revised-98) and 3D-CAM (3-minute diagnostic assessment for CAM-Confusion Assessment Method-defined delirium). In addition to patient assessment, these tests are useful for the clinician in the diagnosis of delirium. The aim of the study is to compare the DRS-R-98 and 3D-CAM tests used in the assessment of POD, and to evaluate their feasibility and the power detecting delirium.

After obtaining ethics committee approval, all patients who undergo orthopedic, urological, general surgery, thoracic and vascular surgery operations in the Istanbul Faculty of Medicine, above 65 years old, with an operation duration longer than 60 minutes will include in this study. Patients who are re-operated, require re-intubation or withdraw their consent will be excluded from the study. This study is planned as an observational, prospective study. Demographic information such as age, gender, height, weight, comorbidities, duration of operation and anesthesia, postoperative pain level, anesthesia and analgesia management, intensive care and hospitalization periods will be recorded from their files. On postoperative day 1, delirium development will be evaluated with DSM-5 diagnostic criteria. All patients will also be evaluated by another physician with both DRS-R-98 and 3D-CAM tests. The same tests will be repeated on postoperative day 2.

ELIGIBILITY:
Inclusion Criteria:

* orthopedic, urological, thoracic, vascular and general surgery operations
* Emergency and elective surgery
* Patients with voluntary consent
* Patients aged ≥ 65 years
* Surgeries longer than 60 minutes

Exclusion Criteria:

* < 65 years old patients
* Operations that take less than 60 minutes
* Patients who do not speak Turkish
* Patients who cannot legally give consent (eg dementia)
* Patients without consent
* Outpatient surgeries
* Reoperated or reintubated patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: ≥ 65 years male and female orthopedic, urological, thoracic, vascular (off-pump) and general surgery operations
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Comparing the tests (3D-CAM and DRS-R-98) in the assessment of postoperative delirium. | 2 days
  the specificity, sensitivity and consistency of 3D-CAM and DRS-R-98 tests used in the evaluation of postoperative delirium. Both tests include sections that assess the patient's responses to the questions asked and also the practitioner's observations

SECONDARY OUTCOMES:
incidence of postoperative delirium | 2 days
  determine the incidence of postoperative delirium
length of hospital stay | 2-21 days
  examine the relationship between delirium and hospital stay
postoperative pain assessment with Numeric Rating Scale (NRS) | 2 days
  Numerical rating scales (NRSs) are the simplest and most commonly used scales.The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."

CONTACTS AND LOCATIONS:
Overall Officials: Zerrin SUNGUR, Prof Dr, Study Chair — Istanbul University Istanbul Faculty of Medicine Department of Anesthesiology and Reanimation
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oh ST, Park JY. Postoperative delirium. Korean J Anesthesiol. 2019 Feb;72(1):4-12. doi: 10.4097/kja.d.18.00073.1. Epub 2018 Aug 24. PMID 30139213
- [Result] Janssen TL, Alberts AR, Hooft L, Mattace-Raso F, Mosk CA, van der Laan L. Prevention of postoperative delirium in elderly patients planned for elective surgery: systematic review and meta-analysis. Clin Interv Aging. 2019 Jun 19;14:1095-1117. doi: 10.2147/CIA.S201323. eCollection 2019. PMID 31354253
- [Result] American Psychiatric Association. Diagnostic and statistical manual of mental disorders (DSM-5Ⓡ). 5th ed. Arlington, American Psychiatric Association Publishing. 2013, pp 596-601.
- [Result] Palihnich K, Inouye SK, Marcantonio ER. The 3D CAM Training Manual for Research. 2014; Boston: Hospital Elder Life Program
- [Result] Cinar MA,Ozmenler KN ,Ozsahin A ,Trzepacz Paula T. Dusunen Adam The Journal of Psychiatry and Neurological Sciences 2014; 3(27): 186-193 DOI: 10.5350/DAJPN2014270301